CLINICAL TRIAL: NCT06316921
Title: Effect of Epidural Patient-controlled Analgesia on Postoperative Pain After Lumbar Spinal Surgeries
Brief Title: Epidural PCA on Pain Relief After L-spine Surgery
Status: Completed | Type: Observational
Sponsor: Taipei City Hospital (Other Government)
Responsible Party: Principal Investigator, Hsin-Chang, Chen, Attending staff of the Department of Orthopedics,, Taipei City Hospital
Other Study IDs: TCHIRB-11003008-E
Record Dates: First submitted 2024-02-23; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Pain, Postoperative; Lumbar Spine Degeneration; Analgesia, Patient-Controlled; Epidural Anesthesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PCA group: Patients received epidural patient-controlled analgesia for postoperative pain.
  Interventions: Procedure: Epidural patient-controlled analgesia
- Control group: Patients received standard of care for postoperative pain.
  Interventions: Procedure: Standard postoperative pain management

INTERVENTIONS:
Procedure: Epidural patient-controlled analgesia — Epidural patient-controlled analgesia for postoperative pain after lumber spine surgery
  Groups: PCA group
Procedure: Standard postoperative pain management — Standard of care for postoperative pain after lumber spine surgery
  Groups: Control group

SUMMARY:
This study aimed to evaluate the effect of epidural patient-controlled analgesia (PCA) on postoperative pain relief after lumbar spine surgeries. The eligible patients received two types of postoperative pain management: PCA and standard pain treatment. Comparisons between the two groups were made in terms of postoperative pain level.

DETAILED DESCRIPTION:
This study included patients who underwent lumbar spine surgeries for degenerative spinal disease. The eligible patients were divided into two groups, the PCA group and the control group, for two types of postoperative pain management. The patients in the PCA group received 72-hour epidural PCA. The PCA catheter was inserted by the surgeon prior to wound closure in the lumbar spine surgery. The PCA catheter was maintained until 72 hours after the surgery and was removed at the postoperative day 4. The control group received postoperative standard pain treatment, including oral acetaminophen and muscle relaxants. No non-steroidal anti-inflammatory drugs were given in this study. All patients were provided the option to request intramuscular morphine injection (0.5 mg of morphine) for additional pain control, with a minimum interval of 6 hours between doses. Pain assessment was conducted using a visual analogue scale on the first four postoperative days and on the day of discharge. At the postoperative day 4, pain assessment was performed before the PCA removal. The level of pain and the number of morphine injections were compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 60 years
2. Having lumbar spine surgeries for degenerative spinal stenosis, spondylolisthesis, herniated intervertebral disc, or osteoporotic spinal fracture with spinal stenosis

Exclusion Criteria:

1. Spinal infection (e.g., tuberculosis, epidural abscess, and vertebral body osteomyelitis
2. Iatrogenic cerebrospinal fluid leakage or dura tear during surgery
3. Spinal tumor or spinal metastasis
4. Having minimally invasive procedures with the bilateral paramedian approach

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent lumbar spine surgeries at Taipei City Hospital
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Pain degree | Postoperative day 1, postoperative day 2, postoperative day 3, postoperative day 4, and the day of discharge (up to 1 month)
  Pain degree was assessed using a visual analogue scale the on the first four postoperative days and on the day of discharge.

SECONDARY OUTCOMES:
The number of morphine injections | The day of discharge (up to 1 month)
  The number of intramuscular morphine injections for additional pain control with a minimum interval of 6 hours between doses.

OTHER OUTCOMES:
Length of hospitalization | The day of discharge (up to 1 month)
  The length of hospital stay (day)
Drainage amount | The day of discharge (up to 1 month)
  The amount of postoperative drainage (ml)

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-chang Chen, MD, Principal Investigator — Taipei City Hospital
Locations (1):
- Taipei City Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No